CLINICAL TRIAL: NCT01642550
Title: A Phase 2, Investigator-Initiated, Randomized, Double-blind, Placebo-controlled Pilot Study to Evaluate the Safety and Efficacy of RM-131 Administered to Females With Anorexia Nervosa
Brief Title: Phase 2 Pilot Study to Evaluate the Safety and Efficacy of RM-131 Administered to Females With Anorexia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Motus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM-131-005
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Anorexia; Eating disorders
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Feeding and Eating Disorders | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RM-131 (Active Comparator): Active study drug - RM-131
  Interventions: Drug: RM-131
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RM-131 — RM-131 (100 mcg) will be administered daily by subcutaneous injection for 28 days.
  Arms: RM-131
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if administration of RM-131 is effective in improving appetite and gastrointestinal symptoms leading to the recovery of patients with anorexia nervosa in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for anorexia nervosa, including weight <85% of ideal body weight (IBW) and amenorrhea for three months;
* Age 18-45 years old;
* Gastrointestinal tract symptoms;
* Non-hormonal method of birth control, which must be used throughout the study. Female patients unable to bear children must have this documented (i.e., tubal ligation, hysterectomy, or post-menopausal, defined as a minimum of one year since the last menstrual period and elevated FSH);
* Stable concomitant medications defined as no changes in regimen for at least 2 weeks prior to baseline;
* Able to provide written informed consent prior to any study procedures and be willing and able to comply with study procedures, including daily SC injections and completion of a daily injection log.
* Patient has a primary care physician or treatment team managing her care.

Exclusion Criteria:

* Use of hormone therapy (including but not limited to estrogen, progesterone) or hormonal methods of birth control (i.e., oral, implantable, or injectable) within eight weeks of screening; or Depo-Provera within six months of screening;
* Pregnancy, lactation or breastfeeding, or a positive serum or urine pregnancy test, within eight weeks of screening;
* History of diabetes mellitus;
* History of purging behaviors greater than once monthly within the last three months;
* Active substance abuse;
* Use of metoclopramide, erythromycin, 5HT3 anti-emetics, or opioid medications within 2 weeks prior to baseline. [Note: these drugs should also not be used post-baseline];
* Hematocrit < 30.0 %, hemoglobin < 10.0 g/dl, potassium < 3.0 mmol/L, fasting glucose > 100 mg/dL, creatinine > 1.5 mg/dL, AST or ALT > 1.5 times the upper limit of normal, or abnormal plasma thyroid stimulating hormone (TSH) level;
* Currently receiving parenteral feeding or enteral feeding, or presence of a nasogastric or other enteral tube for feeding or decompression;
* History of gastric surgery such as fundoplication, gastrectomy, gastric pacemaker placement, vagotomy, bariatric procedure, small or large bowel resection;
* Clinical suspicion, in the opinion of the investigator, of active or symptomatic peptic ulcer disease, cholelithiasis, colitis, celiac sprue, or inflammatory bowel disease;
* Active suicidal ideation;
* Beck Depression Inventory-2 score of ≥ 29;
* Current inpatient hospitalization;
* Allergic or intolerant of egg, milk, wheat or algae, as these are components of the GEBT test meal;
* Participation in a clinical study with an investigational medication or device within the 30 days prior to dosing in the present study;
* Any other reason, which in the opinion of the Investigator, including severe renal, hepatic or cardiac disease, would confound proper interpretation of the study or expose a patient to unacceptable risk.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effect of RM-131 on body weight | Baseline and Day 28
  Change from baseline in body weight.

SECONDARY OUTCOMES:
Effect of RM-131 on gastric emptying time | Baseline and Day 28
  Change from baseline in gastric half-emptying time (t1/2).
Effect of RM-131 on appetite | Baseline and Day 28
  Change from baseline in appetite.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fazeli PK, Lawson EA, Faje AT, Eddy KT, Lee H, Fiedorek FT, Breggia A, Gaal IM, DeSanti R, Klibanski A. Treatment With a Ghrelin Agonist in Outpatient Women With Anorexia Nervosa: A Randomized Clinical Trial. J Clin Psychiatry. 2018 Jan/Feb;79(1):17m11585. doi: 10.4088/JCP.17m11585. PMID 29325236